CLINICAL TRIAL: NCT05774184
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Barzolvolimab (CDX-0159) in Adults With Active Eosinophilic Esophagitis (The "EvolvE" Study)
Brief Title: A Study of CDX-0159 in Patients With Eosinophilic Esophagitis
Acronym: EvolvE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDX0159-08; 2022-001786-12 (EudraCT Number); 2024-512767-30-00 (EU CTIS Number)
Record Dates: First submitted 2023-03-07; First posted 2023-03-17 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Eosinophilic Esophagitis
Keywords: barzolvolimab; esophagitis; EoE; mast cells; CDX-0159
MeSH Terms: conditions — Eosinophilic Esophagitis; Esophagitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Barzolvolimab (CDX-0159) (Active Comparator): 300 mg subcutaneous administration every 4 weeks through week 24
  Interventions: Biological: barzolvolimab
- Placebo then barzolvolimab (CDX-0159) 300mg (Placebo Comparator): Matching placebo subcutaneous administration every 4 weeks through week 16, then 300mg subcutaneous administration every 4 weeks through week 24
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Biological: barzolvolimab — subcutaneous administration
  Arms: Barzolvolimab (CDX-0159)
Drug: Matching Placebo — subcutaneous administration
  Arms: Placebo then barzolvolimab (CDX-0159) 300mg

SUMMARY:
The purpose of this study is to assess the efficacy and safety of barzolvolimab in adult Eosinophilic Esophagitis patients.

DETAILED DESCRIPTION:
The purpose of this study is to assess the efficacy and safety of barzolvolimab in adult Eosinophilic Esophagitis patients.

ELIGIBILITY:
Key Inclusion Criteria

1. ≥ 18 years of age
2. Documented diagnosis of eosinophilic esophagitis (EoE) by endoscopy
3. Peak esophageal intraepithelial eosinophil count (PEC) of ≥ 15 per high power field (hpf) from at least 2 of 3 levels (proximal, mid, and distal) of the esophagus
4. Symptomatic, defined as • Average of ≥ 2 days per week with dysphagia with solid food intake in the 1 month prior to Screening, and • ≥ 4 days with dysphagia within the last 2 weeks prior to randomization
5. On a stable diet which includes solid foods for ≥ 2 months prior to Screening (and throughout the study)
6. Inadequate response to or is inappropriate for and/or intolerant to a standard-of-care treatment for EoE (e.g., PPI, swallowed topical corticosteroids, or dietary elimination)
7. Willing to be compliant with completion of daily questionnaire

Key Exclusion Criteria

1. Diagnosed with hypereosinophilic syndrome or Churg-Strauss syndrome (eosinophilic granulomatosis with polyangiitis)
2. History of clinicopathologic diagnosis of eosinophilic gastritis or eosinophilic duodenitis
3. Known active Helicobacter pylori infection
4. History of coagulation disorders, esophageal varices, achalasia, Crohn's disease, ulcerative colitis, or celiac disease
5. Esophageal dilation within 3 months prior to Screening
6. Prior esophageal or gastric surgery that would confound the assessments of EoE
7. Esophageal stricture that is difficult to pass with a standard adult upper endoscope (9 to 10 mm) or stricture that requires dilation at the Screening EGD
8. Avoiding solid foods or using a feeding tube
9. Regular use of antiplatelet and/or anticoagulant therapy
10. Non-biologic systemic agents within 2 months prior to Screening, including but not limited to corticosteroid (oral, swallowed topical or parenteral), non-steroidal immunosuppressants (e.g., methotrexate, cyclosporin, tacrolimus, mycophenolate mofetil, azathioprine), other immunomodulators (e.g., Jak inhibitors, tyrosine kinase inhibitors), and investigational agents
11. Biologic therapy within 5 half-lives (or detectable serum level) prior to Screening, including but not limited to interleukin (IL)-4 receptor inhibitor (dupilumab), IL-5 inhibitors (e.g., mepolizumab, benralizumab), IL-13 inhibitors (e.g., tralokinumab, lebrikizumab), anti-IgE (e.g., omalizumab), IFN-γ inhibitors, or other approved or investigational biologics
12. Oral immunotherapy (OIT) within 6 months prior to Screening
13. Sublingual immunotherapy (SLIT) and/or subcutaneous immunotherapy (SCIT) Note: Not exclusionary if patient has been on a stable maintenance dose for at least 6 months prior to Screening
14. Receipt of a live vaccine within 2 months prior to the Baseline (Day 1) Visit (patients must agree to avoid live vaccination during study treatment and within 3 months thereafter).
15. Diagnosis of idiopathic anaphylaxis or other severe allergic reactions that in the opinion of the investigator, could increase the patient's risk for systemic hypersensitivity reactions
16. Prior receipt of barzolvolimab

There may be additional criteria your study doctor will review with you to confirm eligibility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2026-01-23 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline to Week 12 in peak intraepithelial mast cell (PMC) count (PMC/hpf). | From baseline to Visit 6 (Week 12)
  Peak esophageal intraepithelial mast cell counts will be determined by counting mast cells in the most inflamed high-power field (hpf) of each of the 3 esophageal (proximal, mid, distal) levels and reported as mast cells/hpf.

SECONDARY OUTCOMES:
Absolute changes from baseline to Week 12 in Dysphagia Symptom Questionnaire (DSQ). | From baseline to Visit 6 (Week 12)
  DSQ is a questionnaire designed to measure difficulty swallowing associated with Eosinophilic Esophagitis (EoE), with total scores ranging from 0 to 84; higher DSQ scores indicate worse symptoms.
Absolute change from baseline to Week 12 in peak intraepithelial mast cell (PMC) count (PMC/hpf) among patients with baseline PMC ≥ 12/hpf. | From baseline to Visit 6 (Week 12)
  Peak esophageal intraepithelial mast cell counts will be determined by counting mast cells in the most inflamed high-power field (hpf) of each of the 3 esophageal (proximal, mid, distal) levels and reported as mast cells/hpf.
Absolute change from baseline to Week 12 in Peak esophageal intraepithelial eosinophil count (PEC) (PEC/hpf). | From baseline to Visit 6 (Week 12)
  Peak esophageal intraepithelial eosinophils will be determined by counting eosinophils in the most inflamed high-power field (hpf) of each of the 3 esophageal (proximal, mid, distal) levels and reported as eosinophils/hpf.
Percent (%) change from baseline to Week 12 in PMC/hpf. | From baseline to Visit 6 (Week 12)
  Peak esophageal intraepithelial mast cell counts will be determined by counting mast cells in the most inflamed high-power field (hpf) of each of the 3 esophageal (proximal, mid, distal) levels and reported as mast cells/hpf.
Incidence of Treatment Emergent Adverse Events. | From first dose through Visit 14 (Week 44)
  The rates of treatment emergent adverse events will be summarized.

CONTACTS AND LOCATIONS:
Locations (45):
- United States (24):
  - AllerVie Clinical Research, Birmingham, Alabama
  - One of a Kind Clinical Research Center, Scottsdale, Arizona
  - GI Alliance- Arizona Digestive Health- Sun City, Sun City, Arizona
  - Del Sol Research Management, LLC, Tucson, Arizona
  - GW Research Inc., Chula Vista, California
  - Connecticut Clinical Research Institute, LLC, Bristol, Connecticut
  - ENCORE Borland Groover Clinical Research, Jacksonville, Florida
  - Gastroenterology of Greater Orlando, Orange City, Florida
  - Treasure Valley Medical Research, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center (KUMC), Kansas City, Kansas
  - Tandem Clinical Research, Marrero, Louisiana
  - Boston Specialists - Boston Food Allergy Center, Boston, Massachusetts
  - NYU Langone Health, New York, New York
  - University of North Carolina (UNC) Hospitals, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - The Clinical Trials Network, LLC, Willoughby, Ohio
  - The Pennsylvania State University (Penn State) Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center-GI Clinical Research Program, Nashville, Tennessee
  - Advanced Research Institute - Ogden, Ogden, Utah
  - Care Access Research, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah
- Australia (3):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - St Vincent's Hospital Melbourne, Melbourne
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - PerCuro Clinical Research Ltd., Victoria, British Columbia
- Germany (3):
  - Universitaetsklinikum Augsburg, Augsburg
  - Klinikum Region Hannover GmbH Burgwedel, Hanover
  - Universitaetsklinikum Magdeburg A.oe.R., Magdeburg
- Italy (5):
  - IRCCS Ospedale San Raffaele, Milan
  - Fondazione Policlinico Universitario A. Gemelli IRCCS - Universita Cattolica del Sacro Cuore, Rome
  - Istituto Clinico Humanitas, Rozzano
  - Azienda Ospedaliera Universitaria OO.RR. San Giovanni di Dio Ruggi d'Aragona-Plesso "Ruggi", Salerno
  - Azienda Ospedaliera - Universitaria Integrata di Verona - Ospedale Borgo Roma, Verona
- Poland (3):
  - Centrum Medyczne Med-Gastr Sp. z o.o., Lodz
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Wojskowy Instytut Medyczny - Panstwowy Instytut Badawczy, Klinika Gastroenterologii i Chorob, Warsaw
- Spain (2):
  - Hospital General Universitario de Alicante Dr. Balmis, Alicante
  - Hospital Clinico San Carlos, Madrid
- United Kingdom (3):
  - St George's Hospital, London
  - St. Thomas' Hospital, London
  - Norfolk and Norwich University Hospital, Norwich

IPD SHARING:
Plan to Share IPD: Undecided